CLINICAL TRIAL: NCT05929209
Title: Exploring Biomarkers in Hereditary Transthyretin Amyloidosis: From Clinical Severity Assessment to New Disease Mechanisms
Brief Title: Exploring Biomarkers in Hereditary Transthyretin Amyloidosis
Acronym: ELBA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Primiano Guido Alessandro, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5470
Record Dates: First submitted 2023-06-07; First posted 2023-07-03 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Hereditary Transthyretin Amyloidosis
Keywords: hereditary transthyretin amyloidosis; neurogenetics; neuromuscular disorders; biomarkers; mitochondrial dysfunction
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Neuromuscular Diseases; Mitochondrial Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment of disease biomarkers (Experimental)
  Interventions: Diagnostic Test: Assessment of disease biomarkers

INTERVENTIONS:
Diagnostic Test: Assessment of disease biomarkers — Assessment of serum, histological and radiological biomarkers

SUMMARY:
Hereditary transthyretin amyloidosis (ATTRv, v for variant) is a severe and heterogeneous systemic condition due to mutations in the transthyretin (TTR) gene.

The availability of disease-modifying therapies has led to an urgent need to have reliable biomarkers capable of assessing the clinical severity of the disease and of monitoring the efficacy of pharmacological treatment. At the same time, early markers for the clinical onset of ATTRv amyloidosis in presymptomatic subjects are needed to enable earlier initiation of anti-amyloid therapy.

In this project the investigators seek to achieve three main goals: to identify and validate disease severity biomarkers in symptomatic patients; to establish disease onset biomarkers of ATTRv amyloidosis in presymptomatic subjects; to explore new pathogenetic mechanisms underlying this multisystem disorder, such as mitochondrial dysfunction and immune response.

DETAILED DESCRIPTION:
Hereditary transthyretin amyloidosis is a severe and heterogeneous systemic condition due to mutations in the transthyretin (TTR) gene. This autosomal-dominant neurogenetic disorder is characterized by an adult-onset with variable penetrance and an extracellular deposition of amyloid in different organs with a prevalent involvement of the somatic and autonomic peripheral nervous system (PNS).

At the same time, the heart, the kidney, the gastro-intestinal system, and the eyes are frequently involved, leading to a lifethreatening multisystem disease with a huge clinical variability and course, and death within 10 years on average. The prevalence of the disease is highly variable between endemic and non-endemic countries and the global prevalence ranges from 5.526 to 38.468. However, the real numbers of ATTRv could even be higher, considering the missing diagnoses and pre-symptomatic carriers regularly followed in each centre. The last few years have been characterized by a significant change in disease management due to a deeper knowledge of the phenotype-genotype correlations and most importantly to the availability of disease-modifying therapies (DMTs). This raises the need for reliable disease biomarkers, in order to monitor the efficacy of the pharmacological treatment and the progression of the disease but also to identify the disease onset in the presymptomatic carriers of TTR gene pathogenic variants.

While enormous progress has been made in diagnostics and treatment in ATTRv, advances in the identification of biomarkers useful for assessing the severity of the disease and the efficacy of pharmacological approaches have not been parallel to this so far. Once molecular diagnosis has been established, ATTRv patients are evaluated in clinical practice and in clinical trials through clinical scales such as the Familial Amyloid Polyneuropathy (FAP) staging system, the Polyneuropathy Disability (PND) score, the Neuropathy Impairment Score (NIS) and its subset, the NIS-lower limbs (NIS-LL) score, and the Norfolk Quality of Life-Diabetic Neuropathy (QoL-DN) questionnaire. However, these purely clinical scales detect a change only when patients have already progressed clinically. It would be desirable to have outcome measures in order to effectively treat presymptomatic patients with a high risk of future clinical worsening.

Furthermore, investigating extraneurological involvement in ATTRv can help identifying disease severity biomarkers and shed light on new general and specific pathogenetic pathways besides those already known. In this context, neurofilament light chain (NfL), a neuronal cytoplasmic protein highly expressed in large calibre myelinated axons, has emerged as a good candidate as a disease biomarker in ATTRv, suggesting a key role in monitoring disease progression.

Providing information about somatic and autonomic small fiber, skin biopsy appears to be a minimally invasive exam able to disclose pathological changes several years before the onset of symptoms. Skeletal muscle can be secondarily involved in ATTRv amyloidosis, as already described for other inherited neuropathies. In this context, muscle MRI can represent a useful tool to evaluate the progression of the pathology.

The main purpose of our study is the definition and validation of disease severity biomarkers in symptomatic patients, able to describe the natural history of the disease and to monitor the efficacy of drug treatments currently available or to be evaluated in future clinical trials. At the same time, the investigators aim to identify measurable criteria capable of early identifying disease onset in presymptomatic subjects. Lastly, the investigators will explore new potentially pathogenetic mechanisms associated with ATTRv, such as mitochondrial dysfunction and the role of inflammation in order to identify a rationale for future innovative therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Molecularly defined patients with hereditary transthyretin amyloidosis, carrying TTR pathogenic variants
2. Presymptomatic carriers of the pathogenic variants in TTR gene
3. Subjects aged 18 years or older
4. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study

Exclusion Criteria:

1. Inability to understand or unwilling to follow the study requirements including attendance at the study center, completion of questionnaires and participation in laboratory testing as called for by the protocol
2. Inability to sign an informed consent
3. Severe psychiatric diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Circulating disease biomarkers in ATTRv amyloidosis | Baseline, weeks 24, 48, 72, 96
  Validation of serum biomarkers of disease (DJ-1, cystatin C, calbindin, uromodulin, GDF-15 and NfL) in patients with ATTRv (baseline assessment).
  Change from baseline in serum levels of disease biomarkers (DJ-1, cystatin C, calbindin, uromodulin, GDF-15 and NfL) at different time points through week 96.
Neuropathological biomarkers in ATTRv amyloidosis | Baseline, week 96
  Baseline assessment of intraepidermal nerve fiber density (IENFD). Change from baseline in intraepidermal nerve fiber density (IENFD) at week 96.
Radiological biomarkers (muscle MRI) in ATTRv amyloidosis | Baseline, week 96
  Baseline assessment of total fatty infiltration score and STIR sequences. Change from baseline in total fatty infiltration score and STIR sequences at week 96.
Circulating disease biomarkers in presymptomatic individuals | Baseline, weeks 24, 48, 72, 96
  Change from baseline in serum levels of disease biomarkers (DJ-1, cystatin C, calbindin, uromodulin, GDF-15 and NfL) at different time points through week 96.
Neuropathological biomarkers in presymptomatic individuals | Baseline, week 96
  Baseline assessment of intraepidermal nerve fiber density (IENFD). Change from baseline in intraepidermal nerve fiber density (IENFD) at week 96.
Radiological biomarkers (muscle MRI) in presymptomatic individuals | Baseline, week 96
  Baseline assessment of total fatty infiltration score and STIR sequences. Change from baseline in total fatty infiltration score and STIR sequences at week 96.

SECONDARY OUTCOMES:
Inflammatory profile in ATTRv amyloidosis | Baseline, week 96
  To document the contribution of inflammation in the ATTRv pathogenesis by assessing serum cytokine levels.
Mitochondrial dysfunction in ATTRv amyloidosis | Baseline
  To document the contribution of mitochondrial dysfunction in the ATTRv pathogenesis by biochemical investigations on serum and muscle/skin.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, ID, Italy